CLINICAL TRIAL: NCT05726149
Title: Efficacy of Unihemispheric Concurrent Dual-Site Anodal Transcranial Direct Current Stimulation Combined With Therapeutic Exercise on Fatigue and Sleep in Fibromyalgia. Randomized Controlled Clinical Trial
Brief Title: UHCDS a-tDCS Combined With Therapeutic Exercise in Fibromyalgia Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Castilla-La Mancha (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UHCDSa-tDCS+EX-Fibromyalgia
Record Dates: First submitted 2023-01-26; First posted 2023-02-13 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Fibromyalgia
Keywords: Neuromodulation; Therapeutic exercise; Fatigue; Sleep
MeSH Terms: conditions — Fibromyalgia; Fatigue | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Real UHCDS a-TDCS + Therapeutic Exercise (Experimental): Real unihemispheric concurrent dual-site anodal transcranial direct current stimulation combined with therapeutic exercise
  Interventions: Device: Real UHCDS a-tDCS; Device: Therapeutic exercise
- Sham UHCDS a-TDCS + Therapeutic Exercise (Sham Comparator): Sham unihemispheric concurrent dual-site anodal transcranial direct current stimulation combined with therapeutic exercise
  Interventions: Device: Therapeutic exercise; Device: Sham UHCDS a-tDCS
- Therapeutic Exercise (Active Comparator): Therapeutic exercise.
  Interventions: Device: Therapeutic exercise

INTERVENTIONS:
Device: Real UHCDS a-tDCS — Real UHCDS a-tDCS (STARTSTIM® 8 stimulator, Neuroelectric Barcelona, Spain) for ten sessions (three sessions per week in weeks 1 and 2; and one session per week in weeks 3, 4, 5 and 6). UHCDS a-tDCS is a galvanic current applied by a cap for 20 minutes at an intensity of 2 milliamps.
  Arms: Real UHCDS a-TDCS + Therapeutic Exercise
Device: Therapeutic exercise — The therapeutic exercise program will include aerobic exercise and muscle strengthening in the same days as UHCDS a-tDCS. The program will last 30-45 minutes.
Device: Sham UHCDS a-tDCS — Sham UHCDS a-tDCS (STARSTIM® 8 stimulator, Neuroelectric Barcelona, Spain) for ten sessions (three sessions per week in weeks 1 and 2; and one session per week in weeks 3, 4, 5 and 6). Sham tDCS will be applied for the same time than real UHCDS a-tDCS.
  Arms: Sham UHCDS a-TDCS + Therapeutic Exercise

SUMMARY:
The purpose of this study is to assess the effects on fatigue and sleep of Unihemispheric Concurrent Dual-Site anodal Transcranial Direct Current Stimulation combined with therapeutic exercise in Fibromyalgia patients.

DETAILED DESCRIPTION:
Fibromyalgia (FM) is one of the rheumatic diseases with the greatest impact on the quality of life, whose etiology and pathophysiology is not yet fully demonstrated.

Perhaps this is why its therapeutic approach is refractory to current treatments.

Apart from the widespread chronic pain characteristic of this syndrome, fatigue is a very disabling symptom in this pathology. It is a complicated, multifactorial, disconcerting and very persistent symptom that is highly frequent in FM. A vast majority of the published studies have focused the symptoms studied in FM on pain, while fatigue and sleep disturbances, despite not being minor symptoms, have not received the same attention.

Neuromodulation treatments with transcranial direct current stimulation (tDCS) have been shown to induce significant analgesia in FM through modification of sensory processing of pain by thalamic inhibitory circuits and improvement of sleep architecture. On the other hand, therapeutic exercise (TE) programs based on aerobic work and global muscle strengthening have been shown to have a beneficial effect in reducing the pain and severity of FM.

None of the four studies conducted so far combining tDCS and TE in fibromyalgia have evaluated the effect on fatigue or sleep. Currently, various studies conclude that Unihemispheric Concurrent Dual-Site anodal Transcranial Direct Current Stimulation (UHCDS a-tDCS) on the dorsolateral prefrontal cortex (DLPFC) and M1 produces a 50% greater modulation of corticospinal excitability. To date, no RCT has studied its effect in subjects with FM.

The present study aims to investigate the effect of UHCDS a-tDCS combined with TE on fatigue and sleep quality in subjects with FM.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years.
* Fulfilled the 2010 American Colleague of Rheumatology criteria for fibromyalgia.
* Able to participated in a therapeutic exercise program.
* Understanding of spoken and written Spanish.

Exclusion Criteria:

* Pregnancy or breastfeeding.
* Metallic implants in the head.
* Tumor, trauma or surgery in the brain.
* Epilepsy or stroke.
* History of substance abuse in the last 6 months.
* Use of carbamazepine in the last 6 months.
* Diagnosed psychiatric pathology.
* Rheumatic pathology not medically controlled.
* Coexisting autoimmune pathology.
* Chronic inflammatory disease (rheumatoid arthritis, erythematosus systemic lupus, inflammatory bowel disease).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Change in fatigue from baseline to post-treatment as assessed by MFI. | Baseline; immediately after intervention; 1-month after intervention
  The version adapted to Spanish from the Multidimensional Fatigue Inventory (MFI) will be used. The scale ranges from 0 to 100. Higher values represent a worse result.
Change in sleep quality from baseline to post-treatment as assessed by MOS-SS. | Baseline; immediately after intervention; 1-month after intervention
  The version adapted to Spanish from the Medical Outcomes Study Sleep Scale (MOS-SS) will be used. The scale ranges from 0 to 100. Higher values represent a worse result.

SECONDARY OUTCOMES:
Fibromyalgia Impact Quality-of-Life | Baseline; immediately after intervention; 1-month after intervention
  It will be measured with the version adapted to the Spanish of the Fibromyalgia Impact Questionnaire (FIQ). The scale ranges from 0 to 100. Higher values represent a worse result.
Blinding | Immediately after intervention.
  Blinding of subjects and researchers will be assessed using the James Index.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Nuestra Señora del Prado, Talavera de la Reina, Toledo, Spain